CLINICAL TRIAL: NCT07237672
Title: Effects of AI Based Physiotherapy on Mandibular Mobility Shoulder Function Whole Body Physical Function Quality of Life and Return to Work in Oral Cancer Patients: 3- and 9-Month Postintervention Follow-Up
Brief Title: AI Based Physiotherapy 3- and 9-Month Follow-Up in Oral Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202412109RIND
Record Dates: First submitted 2025-10-02; First posted 2025-11-20 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Oral Cancer
Keywords: Artificial intelligence; Oral cancer; Maximum interincisal opening; Physical function; Prehabilitation; Physiotherapy
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Masking Description: Follow-up only, no new intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Follow-up) (Experimental): Participants who originally received AI-based physiotherapy will undergo follow-up assessments at 3 and 9 months post-intervention.
  Interventions: Other: AI-based physiotherapy follow-up assessments
- Control group (Follow-up) (Active Comparator): Participants who originally received conventional physiotherapy will undergo follow-up assessments at 3 and 9 months post-intervention.
  Interventions: Other: conventional physiotherapy follow-up assessments

INTERVENTIONS:
Other: AI-based physiotherapy follow-up assessments — AI-based physiotherapy and 3 and 9 months follow-up assessments
  Arms: Experimental group (Follow-up)
Other: conventional physiotherapy follow-up assessments — conventional physiotherapy and 3 and 9 months follow-up assessments
  Arms: Control group (Follow-up)

SUMMARY:
This follow-up clinical study aims to evaluate the sustained effects of two rehabilitation programs (AI-based physiotherapy vs. conventional physiotherapy) for oral cancer patients. Participants who completed the original intervention trial (ClinicalTrials.gov ID: 202411044RINC) will be assessed at 3 and 9 months post-intervention. Outcomes include mandibular mobility, shoulder joint range of motion, functional performance, quality of life, pain, and return-to-work status.

DETAILED DESCRIPTION:
This study is a continuation of our prior trial (ClinicalTrials.gov ID: 202411044RINC), which investigated the short-term effects of AI-based physiotherapy compared with conventional physiotherapy in oral cancer patients.

The current follow-up phase evaluates both groups at 3 and 9 months post-intervention to determine whether initial improvements are maintained and whether they translate into better long-term physical function, quality of life, and return-to-work outcomes. No additional interventions will be delivered; only follow-up assessments are planned.

ELIGIBILITY:
Inclusion Criteria:

* Participants who completed the intervention phase of the previous trial (202411044RINC)
* Age 20-65 years
* Able to attend follow-up assessments at 3 and 9 months

Exclusion Criteria:

* Withdrawal from the original trial
* Cancer recurrence or new cancer-related treatment interfering with functional assessment
* Unable to communicate or comply with follow-up visits

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-12-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand outcome questionnaire | 3 months, 9 months post-intervention
  A total scale from 1 to 100. Higher scores indicate greater disability
EORTC QLQ-C30 questionnaire | 3 months, 9 months post-intervention
  A total scale from 1 to 100. Higher scores indicate greater function

SECONDARY OUTCOMES:
Return-to-work status | 3 months, 9 months post-intervention
  yes/no, time to return, % returned

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Hsia Chen, Ph.D., Principal Investigator — National Taiwan University, College of Medicine
Locations (1):
- School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan, Taipei, Taiwan

REFERENCES:
- [Background] Loos H, Sahm H, Sprenger GA. Glucose-fructose oxidoreductase, a periplasmic enzyme of Zymomonas mobilis, is active in its precursor form. FEMS Microbiol Lett. 1993 Mar 1;107(2-3):293-8. doi: 10.1111/j.1574-6968.1993.tb06045.x. PMID 8472911
- [Background] Baranano CF, Rosenthal EL, Morgan BA, McColloch NL, Magnuson JS. Dynasplint for the management of trismus after treatment of upper aerodigestive tract cancer: a retrospective study. Ear Nose Throat J. 2011 Dec;90(12):584-90. doi: 10.1177/014556131109001209. PMID 22180114
- [Background] Chen CC, Lin CC, Hsieh HP, Fu YC, Chen YJ, Lu TW. In vivo three-dimensional mandibular kinematics and functional point trajectories during temporomandibular activities using 3d fluoroscopy. Dentomaxillofac Radiol. 2021 Feb 1;50(2):20190464. doi: 10.1259/dmfr.20190464. Epub 2020 Aug 12. PMID 32783637
- [Background] Chen SC, Huang BS, Hung TM, Lin CY, Chang YL. Impact of physical and psychosocial dysfunction on return to work in survivors of oral cavity cancer. Psychooncology. 2019 Sep;28(9):1910-1917. doi: 10.1002/pon.5173. Epub 2019 Jul 23. PMID 31291694
- [Background] Chen YH, Liang WA, Lin CR, Huang CY. A randomized controlled trial of scapular exercises with electromyography biofeedback in oral cancer patients with accessory nerve dysfunction. Support Care Cancer. 2022 Oct;30(10):8241-8250. doi: 10.1007/s00520-022-07263-4. Epub 2022 Jul 11. PMID 35821447
- [Background] Chen YH, Huang CY, Liang WA, Lin CR, Chao YH. Effects of Conscious Control of Scapular Orientation in Oral Cancer Survivors With Scapular Dyskinesis: A Randomized Controlled Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211040827. doi: 10.1177/15347354211040827. PMID 34412536
- [Background] Chen YH, Lin CR, Liang WA, Huang CY. Motor control integrated into muscle strengthening exercises has more effects on scapular muscle activities and joint range of motion before initiation of radiotherapy in oral cancer survivors with neck dissection: A randomized controlled trial. PLoS One. 2020 Aug 6;15(8):e0237133. doi: 10.1371/journal.pone.0237133. eCollection 2020. PMID 32760097
- [Background] Chen YH, Liang WA, Hsu CY, Guo SL, Lien SH, Tseng HJ, Chao YH. Functional outcomes and quality of life after a 6-month early intervention program for oral cancer survivors: a single-arm clinical trial. PeerJ. 2018 Feb 21;6:e4419. doi: 10.7717/peerj.4419. eCollection 2018. PMID 29492348
- [Background] Cocks K, Wells JR, Johnson C, Schmidt H, Koller M, Oerlemans S, Velikova G, Pinto M, Tomaszewski KA, Aaronson NK, Exall E, Finbow C, Fitzsimmons D, Grant L, Groenvold M, Tolley C, Wheelwright S, Bottomley A; European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Group. Content validity of the EORTC quality of life questionnaire QLQ-C30 for use in cancer. Eur J Cancer. 2023 Jan;178:128-138. doi: 10.1016/j.ejca.2022.10.026. Epub 2022 Nov 1. PMID 36436330
- [Background] Cohen EE, LaMonte SJ, Erb NL, Beckman KL, Sadeghi N, Hutcheson KA, Stubblefield MD, Abbott DM, Fisher PS, Stein KD, Lyman GH, Pratt-Chapman ML. American Cancer Society Head and Neck Cancer Survivorship Care Guideline. CA Cancer J Clin. 2016 May;66(3):203-39. doi: 10.3322/caac.21343. Epub 2016 Mar 22. PMID 27002678
- [Background] Dijkstra PU, Huisman PM, Roodenburg JL. Criteria for trismus in head and neck oncology. Int J Oral Maxillofac Surg. 2006 Apr;35(4):337-42. doi: 10.1016/j.ijom.2005.08.001. Epub 2005 Nov 8. PMID 16280237
- [Background] Falz R, Bischoff C, Thieme R, Lassing J, Mehdorn M, Stelzner S, Busse M, Gockel I. Effects and duration of exercise-based prehabilitation in surgical therapy of colon and rectal cancer: a systematic review and meta-analysis. J Cancer Res Clin Oncol. 2022 Sep;148(9):2187-2213. doi: 10.1007/s00432-022-04088-w. Epub 2022 Jun 13. PMID 35695931
- [Background] Furtado DA, Pereira AA, Andrade Ade O, Bellomo DP Jr, da Silva MR. A specialized motion capture system for real-time analysis of mandibular movements using infrared cameras. Biomed Eng Online. 2013 Feb 22;12:17. doi: 10.1186/1475-925X-12-17. PMID 23433470
- [Background] Jehn P, Spalthoff S, Lentge F, Zeller AN, Tavassol F, Neuhaus MT, Eckstein FM, Kruskemper G, Gellrich NC, Korn P. Postoperative quality of life and therapy-related impairments of oral cancer in relation to time-distance since treatment. J Cancer Surviv. 2022 Dec;16(6):1366-1378. doi: 10.1007/s11764-021-01118-3. Epub 2021 Oct 5. PMID 34609700
- [Background] Johnson J, Johansson M, Ryden A, Houltz E, Finizia C. Impact of trismus on health-related quality of life and mental health. Head Neck. 2015 Nov;37(11):1672-9. doi: 10.1002/hed.23816. Epub 2015 Jan 27. PMID 24985733
- [Background] Kamstra JI, Reintsema H, Roodenburg JL, Dijkstra PU. Dynasplint Trismus System exercises for trismus secondary to head and neck cancer: a prospective explorative study. Support Care Cancer. 2016 Aug;24(8):3315-23. doi: 10.1007/s00520-016-3131-4. Epub 2016 Mar 8. PMID 26956713
- [Background] Li YH, Chang WC, Chiang TE, Lin CS, Chen YW. Mouth-opening device as a treatment modality in trismus patients with head and neck cancer and oral submucous fibrosis: a prospective study. Clin Oral Investig. 2019 Jan;23(1):469-476. doi: 10.1007/s00784-018-2456-4. Epub 2018 Apr 26. PMID 29696422
- [Background] Loewen I, Jeffery CC, Rieger J, Constantinescu G. Prehabilitation in head and neck cancer patients: a literature review. J Otolaryngol Head Neck Surg. 2021 Jan 6;50(1):2. doi: 10.1186/s40463-020-00486-7. PMID 33407922
- [Background] Marinelli F, Lezcano MF, Alarcon J, Navarro P, Fuentes R. A Novel Technique to Accurately Measure Mouth Opening Using 3D Electromagnetic Articulography. Bioengineering (Basel). 2022 Oct 19;9(10):577. doi: 10.3390/bioengineering9100577. PMID 36290545
- [Background] McMillan H, Barbon CEA, Cardoso R, Sedory A, Buoy S, Porsche C, Savage K, Mayo L, Hutcheson KA. Manual Therapy for Patients With Radiation-Associated Trismus After Head and Neck Cancer. JAMA Otolaryngol Head Neck Surg. 2022 May 1;148(5):418-425. doi: 10.1001/jamaoto.2022.0082. PMID 35297966
- [Background] Michael CM, Lehrer EJ, Schmitz KH, Zaorsky NG. Prehabilitation exercise therapy for cancer: A systematic review and meta-analysis. Cancer Med. 2021 Jul;10(13):4195-4205. doi: 10.1002/cam4.4021. Epub 2021 Jun 10. PMID 34110101
- [Background] Pauli N, Svensson U, Karlsson T, Finizia C. Exercise intervention for the treatment of trismus in head and neck cancer - a prospective two-year follow-up study. Acta Oncol. 2016 Jun;55(6):686-92. doi: 10.3109/0284186X.2015.1133928. Epub 2016 Feb 15. PMID 26878553
- [Background] Shao CH, Chiang CC, Huang TW. Exercise therapy for cancer treatment-induced trismus in patients with head and neck cancer: A systematic review and meta-analysis of randomized controlled trials. Radiother Oncol. 2020 Oct;151:249-255. doi: 10.1016/j.radonc.2020.08.024. Epub 2020 Sep 3. PMID 32890607
- [Background] van der Geer SJ, Reintsema H, Kamstra JI, Roodenburg JLN, Dijkstra PU. The use of stretching devices for treatment of trismus in head and neck cancer patients: a randomized controlled trial. Support Care Cancer. 2020 Jan;28(1):9-11. doi: 10.1007/s00520-019-05075-7. Epub 2019 Nov 7. PMID 31701267
- [Background] Watters AL, Cope S, Keller MN, Padilla M, Enciso R. Prevalence of trismus in patients with head and neck cancer: A systematic review with meta-analysis. Head Neck. 2019 Sep;41(9):3408-3421. doi: 10.1002/hed.25836. Epub 2019 Jun 19. PMID 31215723